CLINICAL TRIAL: NCT03502213
Title: A Prospective Multi-center Observational Trial to Assess Persistence on Active Surveillance When Using the OncotypeDX® Prostate Cancer Assay
Brief Title: Study In Urology Practices Looking At Impact Of OncotypeDX GPS Test On Men Choosing And Remaining On Active Surveillance
Status: Completed | Type: Observational
Sponsor: Genomic Health®, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 09-023
Record Dates: First submitted 2018-03-05; First posted 2018-04-18 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Localized Prostate Cancer; Low Risk Prostate Cancer; Active Surveillance; Active Monitoring; OncotypeDX GPS; Genomic Prostate Score; Genomic Test; Molecular Test
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — fixed paraffin embedded tissue (FFPE) blocks [retained up to 2 years], FFPE sectioned slides [retained up to 2 years], unstained slides [retained up to 2 years], and/or RNA [retained up to 20 years].
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Genomic Health's OncotypeDX® Prostate Cancer Assay is a commercially available laboratory test that measures the activity of certain genes in prostate cancer. The purpose of this study is to better understand how the use of this test result impacts or affects treatment decisions for men newly diagnosed with low risk prostate cancer, their confidence in the treatment decision, and the effects and side effects of the treatment chosen on certain aspects of Quality of Life. This study will also determine what percentage of men choosing an active monitoring program as prescribed by their doctor remain on Active Surveillance and have avoided any treatment at one year after diagnosis after receiving the assay result.

DETAILED DESCRIPTION:
This is a multicenter observational study that evaluates eligible patients who will submit prostate cancer diagnostic biopsy tissues for Oncotype DX Prostate Cancer Assay testing. A physician treatment recommendation will be made and the assay is ordered. The physician will review clinical data, the GPS report and discuss treatment options with the patient. At the following visit, a shared physician-patient treatment decision (immediate treatment or AS) will be made.

Men selecting AS as primary treatment will be followed to assess persistence on AS.

There is no required or standardized AS protocol for this study and the intensity of surveillance will be at the discretion of the investigator. Patients will not be required, but may undergo a standard TRUS guided surveillance biopsy at one year. In this study, the Oncotype DX Prostate Cancer Assay will be assessed on the diagnostic biopsy only and will not be assessed on subsequent biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Clinical stage T1c/T2
* PSA ≤ 20ng/mL
* Biopsy GS ≤ 6 with any number of cores positive, or Biopsy GS 3+4 disease with ≤3 positive cores or ≤ 33% positive cores
* The patient must be ≥ 50 years of age
* The patient must have a life expectancy of > 10 years
* Patient must be able to give consent in English or Spanish

Exclusion Criteria:

* Clinical stage T3a or above
* PSA > 20ng/mL
* Biopsy GS 4+3 or > 8
* Known metastatic prostate cancer
* Positive biopsy for prostate cancer > 3 months ago
* Treatment decision has already been made
* Insufficient tumor in prostate biopsy tissue to perform the assay
* Treatment with androgen deprivation therapy (ADT) prior to prostate biopsy
* Diagnosis made by transurethral resection of prostate (TURP) shavings
* Any psychiatric or psychological conditions
* Contraindications to primary treatment according to physician's judgment

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed with prostate cancer within the last 3 months, with no treatment decision having been made.
Sampling Method: Non-Probability Sample
Enrollment: 489 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Rate of persistence on Active Surveillance at 1 and 2 years after receiving the OncotypeDX Genomic Prostate Score (GPS) | The analysis will estimate the absolute magnitude of the rates of persistence at these two time points (1 and 2 years after receiving GPS)
  The analysis will estimate the absolute magnitude of the rates of persistence at these two time points, and the change between the two rates. The rate of persistence, at the particular timepoint, will be calculated as the proportion of patients who remain on Active Surveillance as of the doctor visit at the time. The rate of persistence will range from 0% to 100%, with 100% indicating all evaluable patients stay on Active Surveillance at the particular timepoint, and 0% indicating no evaluable patient on Active Surveillance.

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-04-24): https://cdn.clinicaltrials.gov/large-docs/13/NCT03502213/Prot_SAP_000.pdf